CLINICAL TRIAL: NCT02946788
Title: An Open Label Study to Document the Treatment Effect of 1 and 2% BPX-01 Minocycline Topical Gel in Moderate to Severe Inflammatory Non-nodular Acne Vulgaris (Protocol Number BPX-01-C04)
Brief Title: Open Label Photo-Documentation Study Of BPX-01 Minocycline Gel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioPharmX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPX-01-C04
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BPX-01 1% (Experimental): BPX-01 1% minocycline topical gel
  Interventions: Drug: Minocycline
- BPX-01 2% (Experimental): BPX-01 2% minocycline topical gel
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — BPX-01 1 or 2% topical gel will be applied to face once daily
  Other Names: BPX-01

SUMMARY:
This is a multi center open label study intended to provide photo documentation and time to response data for BPX-01 1 and 2% minocycline topical gel for the treatment of moderate to severe non-nodular inflammatory acne vulgarism.

DETAILED DESCRIPTION:
This was a 12-week, multi-center, open label, two-arm study. Subjects will be assigned to treatment with 1% or 2% BPX-01 gel. Subjects will apply 1g of the gel as a thin film to the entire face at least 30 minutes before bedtime each night for 12 weeks. Lesion counts, IGA, and Patient-Reported Outcomes (PGI-S and PGI-I) will be performed to assess efficacy. Photographs will be taken to document treatment effect.

Safety will be assessed with the vital signs, brief physical examination, clinical laboratory tests, cutaneous tolerance score, incidence of minocycline-induced skin hyperpigmentation, incidence of visual disturbances and/or headaches suggestive of pseudotumor cerebri, incidence of product related facial staining and collection of adverse events.

ELIGIBILITY:
Inclusion Criteria:

- moderate to severe inflammatory non-nodular acne vulgaris

Exclusion Criteria:

* female subject who is breastfeeding, pregnant or planning a pregnancy during the study
* have other skin condition or disease that would interfere with the study
* have had any prior treatment with minocycline
* have a known or suspected allergy to tetracycline class products
* have used OTC medications for the treatment of facial acne within the last 14 days
* have used any prescription topical or oral medications for the treatment of facial acne in the last 28 days
* have had a facial procedure (chemical peel, dermabrasion, laser, etc) within the last 8 weeks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AnnaMarie Daniels, Study Director — BioPharmX, Inc.
Locations (2):
- United States (2):
  - Study Center, Coral Gables, Florida
  - Study Center, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BPX-01 1%: BPX-01 1% minocycline topical gel
  Minocycline: BPX-01 1 or 2% topical gel will be applied to face once daily before bedtime
- BPX-01 2%: BPX-01 2% minocycline topical gel
  Minocycline: BPX-01 1 or 2% topical gel will be applied to face once daily before bedtime
Period: Overall Study
Arm/Group | BPX-01 1% | BPX-01 2%
Started | 8 | 10
Completed | 8 (October 2017) | 9 (October 2017)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: participants
Groups:
- BPX-01 1%: BPX-01 1% minocycline topical gel
  Minocycline: BPX-01 1 or 2% topical gel will be applied to face once daily at bedtime
- BPX-01 2%: BPX-01 2% minocycline topical gel
  Minocycline: BPX-01 1 or 2% topical gel will be applied to face once daily at bedtime
- Total: Total of all reporting groups
Arm/Group | BPX-01 1% | BPX-01 2% | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — collected at enrollment
  years | 25 [18 to 38] | 25 [18 to 38] | 25 [18 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Inflammatory Lesion Counts at Week 12
Description: difference in number of inflammatory lesions at week 12 as compared to baseline
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: inflammatory lesions
Arm/Group | BPX-01 1% | BPX-01 2%
Number analyzed (Participants) | 8 | 10
inflammatory lesions | 22.3 [10 to 32] | 19.0 [11 to 40]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | BPX-01 1% | BPX-01 2%
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 2/8 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPX-01 1% (N=8) | BPX-01 2% (N=10)
facial redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
facial dryness (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
bloody diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
ear infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
not powered for statistical significance. Small, unblinded study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT02946788/Prot_000.pdf